CLINICAL TRIAL: NCT04120714
Title: Efficacy of Transcranial Direct Current Stimulation (tDCS) in Patients Suffering From Pathological Use of Internet Gaming : Randomized, Controlled, Double-blind, Monocentric Pilot Study
Brief Title: Efficacy of Transcranial Direct Current Stimulation (tDCS) in Patients Suffering From Pathological Use of Internet Gaming
Acronym: StimNET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TROJAK 2019
Record Dates: First submitted 2019-10-08; First posted 2019-10-09 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Pathological Use of Internet Games
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS group (Experimental): Active tDCS
  Interventions: Device: Active tDCS; Other: Questionnaires
- Placebo tDCS group (Placebo Comparator): Inactive tDCS
  Interventions: Device: Placebo tDCS; Other: Questionnaires

INTERVENTIONS:
Device: Active tDCS — active D.C. transcranial stimulation (delivers a low current (1 to 2 mA)) for 10 to 30 minutes, during 5 sessions
  Arms: Active tDCS group
Device: Placebo tDCS — inactive DC transcranial stimulation (delivering a non-significant current at the beginning and end of the stimulation, simulating active stimulation) for 10 to 30 minutes, during 5 sessions
  Arms: Placebo tDCS group
Other: Questionnaires — * visual analogue scale (VAS)
  * impulsivity scale: Barratt Impulsiveness Scale - version 11 (BIS-11)
  * Decision-making scales: Iowa Gambling Task (IGT) and Balloon Analogue Risk Task (BART)
  * Go-No go test
  * HAM-D scale
  * SF-12 quality of life scale

SUMMARY:
The Internet has grown considerably in the last twenty years, and as a result, cases of excessive iinterney use have emerged. These cases, which have clinical similarities with substance addiction, involve the various activities related to the Internet (online gambling, discussion forums, online networking, e-mail, pornography, shopping, etc.). However, to date, only the pathological use of Internet gaming (PUIG) is referenced in the 5th edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5, section III).

In PUIG, an individual loses control when gambling online. He/she typically spends 8 to 10 hours on this activity, sometimes without eating or sleeping. Usual obligations, such as school or work, or family obligations are neglected. PUIG can cause great psychological and social suffering. Neurological complications (epilepsy) and deaths (cardiac arrest) related to PUIG have also been reported. These situations are all the more dramatic because they often affect adolescents and young adults. In Asia, PUIG has become a public health problem. To date, no treatment has been validated for this disorder.

Non-invasive brain stimulation (NIBS) techniques can modulate neural activity in the dorsolateral prefrontal cortex (DLPFC). This modulation makes it possible to reduce addictive behaviours through different mechanisms (reduction of craving, impulsivity, and decision-making disorders). These techniques could be effective for PUIG.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 12 years old
* Patient and/or parents who have given oral consent
* Patient with PUIG (DSM-5 criteria)
* Patient that is motivated and willing to reduce or stop internet gaming

Exclusion Criteria:

* a person who is not affiliated to or not a beneficiary of a social security scheme
* Patient with severe chronic psychiatric comorbidity (schizophrenia, paranoia, chronic hallucinatory psychosis) and bipolar disorder types I and II
* Patient with a gambling addiction
* Patient who has had a recent change (< 1 month) in the prescription of psychotropic treatment
* Patient with an addiction to a psychoactive substance other than tobacco
* Patient receiving psychiatric care without consent or legal protection (guardianship, curatorship)
* Minor patient without parental consent for care
* Patient with severe heart, kidney, liver or lung failure
* Patient with a contraindication to the practice of tDCS: metal parts, medical devices implanted in the brain
* Pregnancy or breastfeeding in progress (negative pregnancy test)
* Patient unable to commit to a three-month follow-up

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Evolution of scores on the IAT scale (Internet Addiction Test) | 4 weeks after tDCS treatment
  Evolution of scores on the IAT (Internet Addiction Test) scale 4 weeks after treatment with tDCS (5 sessions) compared to the 4 weeks preceding brain stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France